CLINICAL TRIAL: NCT07321665
Title: Effects of Physical Activity and Fitness, Cardiovascular- and Psychosocial Health on Medically Assisted Reproduction
Acronym: REPRO-FIT
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: bb25Geiger;2025-00893
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Infertility, Female
Keywords: Medically Assisted Reproduction; Assisted Reproductive Technology (ART); In Vitro Fertilization; Cardiorespiratory Fitness; Cardiovascular Health; Physical Activity; Perceived Stress; Mental Health; Pregnancy Rate
MeSH Terms: conditions — Infertility, Female; Motor Activity; Psychological Well-Being | interventions — Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Health, fitness and lifestyle assessment — Participants undergo a comprehensive, non-interventional longitudinal assessment of physical activity, cardiovascular health, psychosocial factors, sleep quality, and cognitive function integrated into routine medically assisted reproduction care.

SUMMARY:
This prospective observational study aims to investigate the association between physical activity and clinical pregnancy rates in women undergoing medically assisted reproduction. Additionally, it evaluates how cardiorespiratory fitness, cardiovascular health, psychosocial factors, sleep quality, stress, and cognitive function relate to reproductive outcomes.

DETAILED DESCRIPTION:
Infertility affects approximately 8-12% of couples of reproductive age worldwide and represents a major medical and psychosocial burden. Medically assisted reproduction (MAR), including in vitro fertilization (IVF) and intracytoplasmic sperm injection (ICSI), is widely used to address infertility, with more than 12,000 ART cycles performed annually in Switzerland. Despite advances in reproductive medicine, cumulative live birth rates following MAR remain moderate, highlighting the need to better understand modifiable factors that may influence treatment success.

Emerging evidence suggests that general health-related factors-such as physical activity, cardiorespiratory fitness, cardiovascular health, stress, psychosocial well-being, sleep quality, and cognitive function-may play an important role in fertility and MAR outcomes. While moderate physical activity has been associated with improved clinical pregnancy and live birth rates in some studies, the current literature is inconsistent, with conflicting findings regarding the optimal level of activity. Similarly, obesity and cardiovascular risk factors are known to negatively affect fertility and ART outcomes, potentially through mechanisms such as systemic inflammation, insulin resistance, and impaired ovarian responsiveness. Retinal microvascular markers have emerged as early indicators of cardiovascular risk and may provide additional insights into pregnancy-related complications.

Psychological stress, depression, poor sleep quality, and altered psychosocial health are prevalent among women experiencing infertility and may adversely affect reproductive physiology and treatment outcomes. Cognitive and psychosocial factors may further influence fertility indirectly through behavioral, hormonal, and lifestyle pathways. However, these domains are rarely assessed in an integrated and longitudinal manner in women undergoing MAR.

The primary objective of this exploratory, prospective, longitudinal observational study is to examine the association between physical activity and clinical pregnancy rate following MAR in biological women experiencing infertility. Secondary objectives include assessing the relationship of cardiorespiratory fitness, body mass index, blood pressure, retinal microvascular health, psychosocial health, perceived stress, sleep quality, and cognitive function with clinical pregnancy outcomes. Additional objectives are to evaluate short-term changes in physical activity, stress, psychosocial health, sleep, and cognition during hormonal stimulation, as well as changes in retinal microvascular health after completion of the first trimester in cases of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent of the participant has been obtained prior to any screening procedures
* Age 18-43
* Planning to undergo MAR (eg, IUI, IVF, ICSI) - Physically able to cycle for cardiopulmonary exercise testing (CPET)

Exclusion Criteria:

* Any reduction in general state of health preventing from performing hormonal stimulation for MAR
* Absolute and relative contraindications for cardiopulmonary exercise testing (CPET) - No pregnancy at initial screening - Current illicit drug abuse including daily marijuana and CBD consumption (alcohol ≤2 drinks per day allowed)
* Any kind of severe chronic disease (e.g. severe heart failure, active cancer disease)
* Severe renal impairment (e.g. estimated glomerular filtration rate <30 ml/min/m2)
* Known liver cirrhosis or other severe liver impairment
* Uncontrolled dysthyroidism
* Uncontrolled hypertension
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, etc.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women experiencing infertility who are undergoing medically assisted reproduction (MAR) as part of routine clinical care.
Sampling Method: Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate (CPR) after medically assisted reproduction | During the 4 year observational period
  Impact of Physical activity (PA) on clinical pregnancy rate (CPR) following medically assisted reproduction (MAR)

SECONDARY OUTCOMES:
Changes during hormonal stimulation: Physical activity behaviour | preovulatory phase (day 5-14), during hormonal stimulation day (day 31-47), end of first trimester
  Physical activity and inactivity over the past seven days will be assessed using the International Physical Activity Questionnaire (IPAQ).
  Furthermore activity is measured by accelerometer before and during hormonal stimulation.
Changes during hormonal stimulation: Perceived stress | preovulatory phase (day 5-14), during hormonal stimulation day (day 31-47), end of first trimester
  Psychological stress will be assessed using the Perceived Stress Scale.
  The PSS uses a 5-point Likert scale (0-4) for each item, with scores calculated as follows:
  Reverse Scoring: Positive items (e.g., PSS-10: items 4, 5, 7, 8) are reverse-scored (0 = 4, 1 = 3, 2 = 2, 3 = 1, 4 = 0).
  Total Score: Sum all item scores after reversing positive items. PSS-10: Range 0-40
  Interpretation: Higher scores indicate greater perceived stress. General guidelines (not diagnostic) include:
  PSS-10: 0-13 (low), 14-26 (moderate), 27-40 (high)
Changes during hormonal stimulation: Depressive symptoms | preovulatory phase (day 5-14), during hormonal stimulation day (day 31-47), end of first trimester
  Depressive symptoms will be assessed using the Patient Health Questionnaires-9 (PHQ-9).
  Scoring: Each question is scored 0 (not at all) to 3 (nearly every day), with a total score up to 27.
  Severity Levels:
  0-4: Minimal depression 5-9: Mild 10-14: Moderate 15-19: Moderately severe 20-27: Severe.
Changes during hormonal stimulation: Anxiety symptoms | preovulatory phase (day 5-14), during hormonal stimulation day (day 31-47), end of first trimester
  Anxiety symptoms will be assessed using the Generalized Anxiety Disorder-7 questionnaire (GAD-7).
  Each answer is 0 (not at all), 1 (several days), 2 (more than half the days), or 3 (nearly every day).
  Total Score (0-21): Sum of all 7 items.
  Severity Levels:
  0-4: Minimal anxiety. 5-9: Mild anxiety. 10-14: Moderate anxiety. 15-21: Severe anxiety.
Changes during hormonal stimulation: Body image | preovulatory phase (day 5-14), during hormonal stimulation day (day 31-47), end of first trimester
  Body image will be assessed using the Body Appreciation Scale-2 (BAS-2). Body Appreciation Scale-2 (BAS-2) is a 10-item measure of one's acceptance, favorable opinions and respect of their own body.
  Response Options:
  Never - 1 Seldom - 2 Sometimes - 3 Often - 5 Always - 5
  Scoring Procedures The mean of the 10 items is calculated for the total score. Higher scores indicate higher body appreciation.
Changes during hormonal stimulation: Sleep quality | preovulatory phase (day 5-14), during hormonal stimulation day (day 31-47), end of first trimester
  Sleep disturbances will be assessed using the Insomnia Severity Index (ISI). The Insomnia Severity Index (ISI) uses a 0-28 scale, with each of its seven items rated 0 (none) to 4 (very severe), where higher scores mean worse insomnia, categorizing results into no insomnia (0-7), subthreshold (8-14), moderate (15-21), and severe (22-28) insomnia, indicating clinical significance and potential need for treatment as scores rise
Changes during hormonal stimulation: Quality of life | preovulatory phase (day 5-14), during hormonal stimulation day (day 31-47), end of first trimester
  Quality of life will be assessed using the WHO-5 Well-Being Index. The WHO-5 Well-Being Index scaling uses a 6-point Likert scale (0 to 5) for five questions about the past two weeks, summing them for a raw score (0-25), then multiplying by 4 to get a final score (0-100), where 0 is worst and 100 is best; scores below 50 suggest poor well-being and potential depression needing further checks, with a score of 28 or below often indicating depression
Changes during hormonal stimulation: Cognitive function | preovulatory phase (day 5-14), during hormonal stimulation day (day 31-47), end of first trimester
  Cognitive function will be tested by strooper task.
Changes during hormonal stimulation: Nutrition | preovulatory phase (day 5-14), during hormonal stimulation day (day 31-47), end of first trimester
  Dietary habits will be screened by mini-EAT (Eating Assessment Tool). Mini-Eating Assessment Tool (Mini-EAT) is a 9-item rapid dietary screener that includes fruits/vegetables, whole grains, refined grains, fish/seafood, legumes/nuts/seeds, low-fat dairy, high-fat dairy, and sweets consumption.
Amount and type of gonadotropins used | During the 4 year observational period
Ovulation trigger medication | During the 4 year observational period
Amount of eggs collected per ovarian pick-up (OPU) | During the 4 year observational period
Complications (Ovarian hyperstimulation syndrome, ovarian torsion, bleeding or infection after OPU) | During the 4 year observational period
IVF fertilisation rate | During the 4 year observational period
ICSI fertilisation rate | During the 4 year observational period
Blastocyst development rate | During the 4 year observational period
Blastocyst grading | During the 4 year observational period
Evaluation of fresh vs. frozen embryo transfer | During the 4 year observational period
Implantation rate | During the 4 year observational period
Time to pregnancy | During the 4 year observational period
Miscarriage rate (before twelve weeks of pregnancy) | During the 4 year observational period
Pregnancy complications | During the 4 year observational period
Preterm birth | During the 4 year observational period
Cumulative life birth rate | During the 4 year observational period
Fetal malformations | During the 4 year observational period
Perinatal death | During the 4 year observational period

CONTACTS AND LOCATIONS:
Overall Officials: James Geiger, Study Chair — University Hospital of Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland